CLINICAL TRIAL: NCT03903601
Title: Concentration of Trimethylamine Oxide (TMAO) in Blood Plasma as a Risk Factor for Vascular Cerebral Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Robert Olek, Associate Professor, Gdansk University of Physical Education and Sport
Other Study IDs: DSRiK/10/2019
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-02

CONDITIONS: Vascular Diseases; Leukoaraiosis; Ischemia, Cerebral
Keywords: trimethylamine-N-oxide; magnetic resonance imaging; cognitive functions
MeSH Terms: conditions — Vascular Diseases; Leukoaraiosis; Brain Ischemia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic changes: Patients with ischemic changes in the brain diagnosed by MRI
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Blood samples collection; Diagnostic Test: Neuropsychological tests
- No ischemic changes: Patients without ischemic changes in the brain diagnosed by MRI
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Blood samples collection; Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) to diagnose ischemic changes in the brain.
Diagnostic Test: Blood samples collection — Trimethylamine N-oxide (TMAO) concentration, oxidative stress markers and endothelial dysfunction markers will be determined in blood samples.
Diagnostic Test: Neuropsychological tests — Cognitive functions assessment

SUMMARY:
The primary aim of the current research project is to answer the question, whether plasma trimethylamine N-oxide (TMAO) level may be used as a marker of ischemic changes in the brain. TMAO is associated with endothelial dysfunction, inflammation and oxidative stress.

The hypothesis is that circulating TMAO level may predict leukoaraiosis (LA) and/or stroke.

Secondary, the investigators would like to examine whether plasma TMAO concentration is related to cognitive impairment and determine whether choline consumption is associated with an incidence of LA severity and dementia.

DETAILED DESCRIPTION:
In the study, subjects will be recruited in the hospital among the patients with brain MRI performed within past 4 weeks. All MRI scans will be reviewed by the neurologist to evaluate ischemic changes. Upon detection of LA, patients (n=150) will be informed about the study aims. In the same time, aged- and sex-matched control group (n=150) with no detected ischemic changes will be recruited.

In each group, the blood samples will be collected, to determine the concentration of plasma TMAO, oxidative stress markers, as well as serum endothelial dysfunction markers and biochemical parameters. To determine the cognitive performance psychological test will be carried out. The diet of all recruited participants, with special consideration on the choline-rich products and supplements, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* the ischemic changes in the brain (diagnosed by neurologist by MRI scans)

Exclusion Criteria:

* no ischemic changes in the brain (diagnosed by neurologist by MRI scans)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from 7th Navy Hospital in Gdansk, which had a brain MRI performed within the past 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Brain Magnetic Resonance Imaging (MRI) | before qualifying for the study, during the recruitment period
  Leukoaraiosis severity will be evaluated in MRI scans according to the Fazekas' scale. Will be grading scale for periventricular hyperintensities (PVH) and scale of deep white matter hyperintensities.
Trimethylamine-N-oxide (TMAO) blood concentration | up to 4 weeks after brain MRI
  TMAO concentration determined by the ultra-performance liquid-chromatography tandem mass spectrometry (UPLC-MS/MS), marked in µmol/l.

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor (BDNF) | up to 4 weeks after brain MRI
  BDNF concentration determined in serum by ELISA method, marked in pg/mg.
Mini Mental State Examination (MMSE) | up to 4 weeks after brain MRI
  MMSE is a screening tool for cognitive functions impairment.
Trail Making Test (TMT) | up to 4 weeks after brain MRI
  TMT test to determine the executive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, PhD, Principal Investigator — Gdansk University of Physical Education and Sport
Locations (1):
- University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland